CLINICAL TRIAL: NCT02170324
Title: GLP-1 Agonism Stimulates Browning of Subcutaneous White Adipose Tissue in Obesity Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinology Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014Wze091
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 agonism group (Experimental): Exenatide injection 10 ug twice daily for 10 days subcutaneously.
  Interventions: Drug: Exenatide
- Placebo group (Placebo Comparator): 0.9 % sodium choride 0.1 ml twice daily for 10 days subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide
  Arms: GLP-1 agonism group
Drug: Placebo
  Arms: Placebo group

SUMMARY:
Adipose tissues, which include white adipose tissue (WAT) and brown adipose tissue (BAT), play an essential role in regulating whole-body energy homeostasis. Excess expansion of WAT due to positive energy balance and defects in thermogenic gene expression in BAT are associated with obesity and various metabolic diseases. Until 2009 the question of whether adult humans had BAT and whether it could conceivably contribute to whole body energy usage in a meaningful way was a matter of vigorous debate. The publication of three apppers in the New England Journal of Medicine that demonstrated adult humans do have BAT, that it can be activated, and that this activation appears to be defective in obesity reframed the debate, and revived interest in BAT physiology. Recent studies also reveal the presence of a subset of cells in WAT that could be induced by environmental or hormonal factors to become ''brown-like'' cells, and this ''beigeing'' process has been suggested to have strong antiobesity and antidiabetic benefits.

The extrapancreatic actions of glucagon-like peptide-1 (GLP-1) on endothelial cells and the liver have been reported. Additionally, effects of GLP-1 on adipose tissue have been described. Studies performed in isolated adipocytes have demonstrated that GLP-1 has the ability to induce both lipogenic and lipolytic mechanisms in white adipose tissue (WAT) . More recent study showed that GLP-1 agonism stimulates brown adipose tissue thermogenesis and browning through hypothalamic AMP-activated protein kinase (AMPK) in animal. However, there is no data clearly show that GLP-1 agonism stimulates browning of subcutaneous white adipose tissue (SWAT) in human obesity.

DETAILED DESCRIPTION:
Individuals were treated for 10 days. Biopsy for subcutaneous white adipose (1.5X1.5X1.5cm) was performed before and after 10 days treatment programme under local anesthesia. Measure the brown fat characteristics of biopsy samples.The sample was immediately processed in 3 sections.One part was stored for immunohistology and western blot, the second was snap-frozen for estimation of biochemical markers, and the remainder was used to harvest small subcutaneous arteries with micro-dissection. Also, the perivascular adipose tissue (PVAT) was studied on the changes of morphology and possible signal pathways before and after GLP-1 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 30 kg/m2
* Men
* Age 20 - 30 years old

Exclusion Criteria:

* BMI < 30 kg/m2
* Diabetes
* Hypertension
* Use of medicines

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The expression of brown adipose related genes in subcutaneous white adipose tissue | 3 months
  Brown fat characteristics of biopsy samples will be assessed by determining the expression levels of uncoupling protein-1 (UCP-1), peroxisome proliferator-activated receptor (PPAR)-r, peroxisome proliferator-activated receptor r coactivator 1 a (PGC1a) , growth factor receptor binding protein-10 (Grb10), PR domain containing 16 (PRDM16); In addition, a combination of PET and computed tomography (CT) - with the glucose analogue 18F-fluorodeoxyglucose (18F-FDG) as a tracer will be performed for brown adipose tissue before and after GLP-1 agonism treatment programme.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China